CLINICAL TRIAL: NCT01726868
Title: Clinical Study to Evaluate the Efficacy of Blood Purification Therapy on Cholesterol Crystal Embolism
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Japan Community Health Care Organization Sendai Hospital (Other)
Responsible Party: Principal Investigator, TOSHINOBU SATO, MD, PhD, Japan Community Health Care Organization Sendai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCE-001
Record Dates: First submitted 2012-11-10; First posted 2012-11-15 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Cholesterol Embolism
MeSH Terms: conditions — Embolism, Cholesterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liposorber LA-15 System (Experimental)
  Interventions: Device: Liposorber LA-15 System

INTERVENTIONS:
Device: Liposorber LA-15 System — Six sessions of blood purification treatment with Liposorber LA-15 System.

SUMMARY:
The aim of this study is to evaluate efficacy and safety of blood purification therapy on renal dysfunction by cholesterol crystal embolism.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria.

* Patients who had cardiac catheterization or vascular surgery in the last 24 weeks before the time of obtaining informed consent.
* Patients who satisfy all of the following criteria or are diagnosed as CCE by skin or renal biopsy.

  1. Patients with progressive renal dysfunction in the course of weeks or months.
  2. Patients with skin lesions such as livedo reticularis of lower extremities or blue toe syndrome.
  3. Eosinophil count is more than 400 per microliter.
* Patients who or patients whose legal representative understood the requirements of the study and signed the informed consent forms.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded.

* Patients with contraindication to anticoagulant (Nafamostat Mesilate).
* Blood purification therapy is inapplicable because of severe heart failure, acute myocardial infarction, severe arrhythmia, acute stroke, or severe uncontrollable hypertension or hypotension.
* Patients with body weight less than 40kg.
* Patients with a history of allergic reaction or hypersensitivity to blood purification.
* Patients who cannot stop taking ACE inhibitors.
* Patients with any disease in which corticosteroid, statin are contraindicated.
* Patients participated in another clinical trial or study at the time of obtaining informed consent.
* Patients receiving chronic hemodialysis.
* Otherwise, patients who are judged by the investigator as being unsuitable for inclusion in the study.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2013-07; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic hemodialysis | Six months

SECONDARY OUTCOMES:
Dose of drugs | Six months
Incidence of lower limb amputation | Six months
Incidence of gangrene | Six months
Incidence of multi organ failure | Six months
Survival rate | Six months
Incidence of adverse events | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Toshinobu Sato, MD, PhD, Study Director — Japan Community Health Care Organization Sendai Hospital
Locations (1):
- Sendai Shakaihoken Hospital, Sendai, Miyagi, Japan

REFERENCES:
- [Derived] Ishiyama K, Sato T. Efficacy of LDL apheresis for the treatment of cholesterol crystal embolism: A prospective, controlled study. Ther Apher Dial. 2022 Apr;26(2):456-464. doi: 10.1111/1744-9987.13706. Epub 2021 Jul 11. PMID 34216189